CLINICAL TRIAL: NCT03398044
Title: Administration of Dexamethasone in PONV Prophylaxis in Children Between 3 and 15 Years of Age Undergoing Adenotomy in General Anaesthesia; Risks and Side Effects of the Treatment
Brief Title: Administration of Dexamethasone in PONV Prophylaxis in Children Undergoing Adenotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FNO-KARIM-5
Record Dates: First submitted 2018-01-05; First posted 2018-01-12 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Nasal Obstruction; Nasopharyngeal Obstruction; Snoring; Apnea, Obstructive; Hearing Loss; Otitis
MeSH Terms: conditions — Nasal Obstruction; Snoring; Sleep Apnea, Obstructive; Hearing Loss; Otitis | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: The study subjects were randomised into two arms, one group with active treatment using dexamethasone, and the other arm of subjects receiving placebo.
Who Masked: Participant, Investigator
Masking Description: Masking was provided by a nurse not participating upon the research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone (Experimental): Patients randomised into the Dexamethasone arm will be administered active studied drug during anaesthesia induction.
  Interventions: Drug: Dexamethasone
- Placebo (Placebo Comparator): Patients randomised into the control Placeboarm will be administered placebo during anaesthesia induction.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone will be administered to patients randomised into the active treatment arm, in order to determine the influence upon PONV incidence.
  Arms: Dexamethasone
Drug: Placebo — Placebo will be administered to patients randomised into the control group arm.
  Arms: Placebo

SUMMARY:
Adenotomy, together with tonsillectomy, belongs among the most frequently performed surgical procedures in paediatric patients. These surgical procedures are associated with the second highest incidence of post-operative nausea and vomiting (PONV) (following strabism correction surgery) in paediatric surgery. PONV is associated, apart from the discomfort for the child, with a number of complications: dehydration, metabolic disruption or danger of haemorrhage and aspiration of the gastric content. Adenotomy is a typologically completely different surgical procedure, with a different target structure of the surgery, and the length and invasiveness of the procedure. Thus, it is possible to expect a difference in PONV incidence when compared to tonsillectomy. Adenotomy is a surgical procedure performed namely in children of the pre-school age. This is associated, among others, also with the problem of objectivization of post-operative nausea, which is very difficult to verbalize in small children, being a subjective feeling of body discomfort. It is possible to expect that the overall incidence of PONV will be significantly underestimated.

DETAILED DESCRIPTION:
Randomization The study subjects were randomized into two arms, using computer-generated sequence of binary code: interventional arm with dexamethasone administration and control group with a placebo - physiological solution. Anaesthesiology nurse, who was not a part of the research team, randomly selected a vial for each enrolled patient, which was later administered to the patient. The number of the ampule corresponded with the patient's number.

Standardized anaesthesiology protocol General anaesthesia was administered in every paediatric patient according to a standardized anaesthesiology protocol. Each subject received premedication with midazolam in the dose of 0.5 mg/kg of body weight, per orally, 45 minutes before the surgical procedure. Inhalation induction of general anaesthesia was initiated with Sevoflurane, the vaporizer was set to 8%, using the carrying mixture of gases O2/air in the 1:1 ratio. After induction of anaesthesia, peripheral venous line was secured, with subsequent administration of an opioid - Sufentanil in the dose of 0.2 uq/kg of body weight, together with the research drug in the dose of 0.15mg/kg of body weight, with the maximum dose of 4 mg administered intravenously. The airways were secured in accordance with standard procedures used at our centre - armed laryngeal mask. In case of any leakages, air leaks, or any other problems with the laryngeal mask, the airways were secured with orotracheal intubation and introduction of tamponade into hypopharynx. General anaesthesia was further maintained using Sevoflurane, towards the values of MAC 1.2-1.5. Fluid therapy was guided by the 4/2/1 ml/kg of body weight /hr. rule - using Ringer's solution. Each subject was given standard analgetization for the early post-operative period: Paracetamol in the dose of 15mg/kg of body weight i.v. in the course of 10 minutes of the surgical procedure. Standard monitoring was provided for every patient: ECG, measurement of blood pressure, saturation, capnometry, inspiration and expiration Sevoflurane concentrations. After the surgery, every patient was woken up from anaesthesia, the laryngeal mask was removed (extubation) with spontaneous ventilation, the patient was further transferred to PACU.

Data collection Anaesthesiology team (anaesthetist + nurse), who was responsible for administration of general anaesthesia according to the standardized protocol, and who was trained to perform the study according to the study protocol, recorded the data concerning Dexamethasone/Placebo administration into a special Case Report Form, containing identification and number of the study drug. The form was transferred together with the patient to PACU, where the occurrence of PONV was monitored and recorded, together with the first value of the BARF score, by a PACU nurse and the child's parent. The form concerning the incidence PONV at inpatient department was provided for the parent who was present at the bedside of the patient at all times, up to the child's discharge from the hospital - the parent noted the number of vomiting episodes and BARF score 8 hours after the surgery (late BARF score); the parent was further instructed to ask the child ever 2 hours about possible sickness. In case of vomiting, the time and number of vomiting episodes were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age (3-15 years)
* Signed informed consent by legal representatives of the child and patients (depending on the patient's age)
* Patients indicated for surgical procedure: adenotomy

Exclusion Criteria:

* ASA III and more
* Chronic medication: corticosteroids
* Malignant disease

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
PONV incidence | 24 months
  To determine, whether Dexamethasone administered in single prophylactic dose of 0.15mg/kg of body weight of the child, after general anaesthesia induction, statistically significantly decreases the incidence of PONV in paediatric patients at the age between 3 and 15 undergoing adenotomy

SECONDARY OUTCOMES:
Nausea incidence | 24 months
  To assess the incidence of nausea in children using BARF score and monitoring of possible difference between the interventional and control groups

CONTACTS AND LOCATIONS:
Overall Officials: Michal Frelich, MD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No